CLINICAL TRIAL: NCT02287051
Title: Acceptance and Compliance of Split-dose Bowel Preparation for Colonoscopy in Clinical Practice
Brief Title: Bowel Prep Acceptance in Clinical Practice
Status: Completed | Type: Observational
Sponsor: Valduce Hospital (Other)
Responsible Party: Principal Investigator, Arnaldo Amato, MD, Valduce Hospital
Other Study IDs: 7/14
Record Dates: First submitted 2014-10-12; First posted 2014-11-10 (Estimated); Last update posted 2014-11-10 (Estimated); Status verified 2014-11

CONDITIONS: Colonoscopy: Bowel Preparation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- colonoscopy population

SUMMARY:
Bowel preparation for colonoscopy is crucial, since the diagnostic accuracy of the procedure depends on an adequate visualization of the mucosa of the colon.There is strong evidence that the quality of bowel preparation is inversely correlated with the interval between the end of the assumption of the purgative and the start of colonoscopy (shorter intervals are associated with higher levels of preparation).Recent studies have shown that split dose prep significantly improves the quality of bowel cleansing. In light of these data, both the American College of Gastroenterology (ACG) and the European Society of Gastrointestinal Endoscopy (ESGE) recommend now split dose prep in order to improve the quality of bowel cleansing. Despite these recommendations, the uptake of schemes in divided doses appears clearly underused in actual clinical practice. In particular, in Italy only a few centers routinely adopt the regime split as their first choice for the preparation for colonoscopy.The reasons why the "split dose" is under-utilized in clinical practice are not entirely clear, but probably in part reflecting gastroenterologists' concerns about potential elements that theoretically could make it less acceptable to the patient (get up early in the morning, potential problems during the journey from home to the hospital) The hypothesis of the study is that many patients would still be willing to accept these potential drawbacks if they were adequately informed about the positive impact of the scheme in divided doses on the effectiveness of bowel preparation, which results in higher reliability of the examination, shorter duration of the procedure, and less risk of rescheduling the exam in the near future

ELIGIBILITY:
Inclusion Criteria:

* adult patientes undergoing colonscopy

Exclusion Criteria:

* afternoon colonoscopy
* partial colonoscopy
* ASA III-IV
* pregnancy
* incapacity to give informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: population undergoing colonoscopy
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2014-03; Primary Completion 2014-06 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
acceptance | 3 month
  structured questionnaire on acceptability and problems related to the modality of the preparation
compliance | 3 month
  structured questionnaire on completeness and difficulties related to the modality of the preparation

REFERENCES:
- [Derived] Radaelli F, Paggi S, Repici A, Gullotti G, Cesaro P, Rotondano G, Cugia L, Trovato C, Spada C, Fuccio L, Occhipinti P, Pace F, Fabbri C, Buda A, Manes G, Feliciangeli G, Manno M, Barresi L, Anderloni A, Dulbecco P, Rogai F, Amato A, Senore C, Hassan C. Barriers against split-dose bowel preparation for colonoscopy. Gut. 2017 Aug;66(8):1428-1433. doi: 10.1136/gutjnl-2015-311049. Epub 2016 Apr 19. PMID 27196589